CLINICAL TRIAL: NCT05461521
Title: Post-traumatic Stress Disorder in Relatives of Patients Admitted to the ICU: a Multicenter, Observational, Prospective Study (FAME Observational)
Brief Title: Improving FAMily Members' Experience in the ICU
Acronym: FAME
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RC22_0078
Record Dates: First submitted 2022-07-04; First posted 2022-07-18 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Stress Disorders, Post-Traumatic; Family Members
Keywords: Family Members of a Patient Hospitalized in Intensive Care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Objective: to identify biomarkers of PTSD in family members of patients admitted to the ICU
  * Number of family members: 350
  * Samples : 4 blood tubes (for DNA, RNA and plasma): total of 19 ml.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Family members of patients admitted to the ICU
  Interventions: Other: Family members of patients admitted to the ICU
- Health care professionals
  Interventions: Other: Health care professionals
- Patients
  Interventions: Other: Patients

INTERVENTIONS:
Other: Family members of patients admitted to the ICU — At inclusion:
  * Collection of demographic data, Anxiety-Depression Scale (HADS), Insomnia Severity Index (ISI), Resilience Insomnia Severity Index (ISI), Resilience Scale (CD RISC 10), Peritraumatic Dissociation Peritraumatic Dissociation Experience Scale (PDEQ) and MEDEC questionnaire.
  * Venous blood sampling at 350 relatives
  * Upon discharge of the patient (alive or deceased): Resuscitation questionnaire, HADS, ISI and PDEQ.
    3 months after discharge: Demographic questionnaire, Post Traumatic Stress Disorder questionnaire (PCL-5), THS Past Trauma Experience Questionnaire, HADS experiences, HADS, ISI, CD RISC 10, MEDEC and Who- assist questionnaire (Question 2) on the use of psychoactive substances.
    6 months after patient discharge: PCL-5, HADS, ISI, CD RISC 10, MEDEC, Who-assist (Question 2) and Prolonged Grief disorder (PG-13) questionnaire on bereavement if patient died in the ICU.
  Groups: Family members of patients admitted to the ICU
Other: Health care professionals — All professionals in all categories and in all participating departments will be asked to complete questionnaires to assess the level of conflict, work stress and burn out in the units : Masclach Burnout Inventory (MBI), Job Content Questionnaire (JCQ), Ethical Decision-Making Climate Questionnaire (EDMCQ), Professional Quality Of Life scale (ProQOL), Connor-Davidson Resilience scale (CD-RISC 10), Cultural Awareness Scale (CAS).
  Groups: Health care professionals
Other: Patients — Inclusion (at D3 after admission to the ICU): collection of demographic data Discharge from the ICU: characteristics of the stay and outcome (alive/deceased)
  Groups: Patients

SUMMARY:
The aim of the present research is to set up a large multicentric, prospective cohort of family members of patients admitted to intensive care. The data collected will concern the patients and their family members, the caregivers and the functioning of the services during the collection period. This cohort will allow:

1. to carry out a quantitative evaluation of post-traumatic stress disorder (PTSD) in a large number of family members, to determine the risk factors in relation to the characteristics of the family members, and to define a predictive model of PTSD in this population
2. to determine the factors related to the operating conditions of the resuscitation services that favor the occurrence of PTSD in the family members,
3. to create a biological bank from blood samples taken from family members,
4. to carry out a qualitative study allowing a psychological and sociological analysis of the experience of the family members concerning the hospitalization in intensive care of their loved one.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* ≥18 years old
* Treated in the ICU with invasive mechanical ventilation for 48 hours
* Having been visited by at least one family member within 72 hours of the 48th hour of intubation in intensive care
* Having been informed of the study and not having objected to the use of their medical medical data prior to discharge from the ICU if they are able to receive the information the information at the time of inclusion or consent of the family member obtained for the inclusion of the patient if the patient is not able to do so at the time of at the time of inclusion

Family members :

* ≥18 years old
* Identified if possible by the patient as the person to be referred or to be informed, or, in the case of a patient unable to express him/herself, identified by the caregivers as the "patient's close referent".
* Understanding and speaking French
* Having been informed of the study and having consented to participate in it during a visit of the patient
* Inclusion between H48 and H120 post-intubation of the patient in the ICU (if the patient is still intubated at the time of inclusion)
* Having given their telephone number
* Being covered by a social security plan.
* Only one relative of the patient is included in the study Service Professionals: All professionals in all categories and in all participating participating services who have been informed of the study and have consented to participate.

Exclusion Criteria:

Patients:

* No family member or no family member visit
* No consent to participate from family member
* Organ donation planned or contemplated
* Pregnant or parturient woman
* Detained or deprived of liberty
* Under guardianship or curator
* No social security

Family members :

* Social context making follow-up and telephone interviews difficult (homeless, not residing in Europe or in the DOM)
* Inability to give a "stable" personal cell phone number
* Under guardianship or curator
* Unable to communicate on the phone (hearing impairment...)

Service Professionals:

* Not on duty (locum tenens or interim team, only on-call) on call)
* Not qualified (Physician: at least intern, nurse DE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family members : 1346 family members of 1346 patients admitted to the ICU and treated with invasive mechanical ventilation will be included in the research. Only one person among the patient's family members will be concerned by the study. The inclusion window will be 72 hours, starting from the 48th hour after the patient's intubation in the ICU and ending at the 120th hour after intubation.
  Patients: 1346 patients treated with invasive mechanical ventilation will be included in this research. Information about the study will be given to the patient at the same time as to the family member if the patient is conscious, or as soon he is able to receive the information.
  Caregivers: All professionals in all categories and in all participating departments will be asked to complete questionnaires to assess the level of stress and burn out in the units. Participation in the study will be participation in the study will be offered to them at the beginning of the study in the department.
Sampling Method: Probability Sample
Enrollment: 1346 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
To determine the factors associated with post-traumatic stress disorder (PTSD) in family members of patients admitted to the ICU, and. | at 3 months after the patient's discharge from the ICU
  The primary endpoint is the proportion of family members who developed PTSD 3 months after the patient's discharge from the ICU assessed by the Post-traumatic stress disorder CheckList (PCL-5) version Diagnostic and Statistical Manual of Mental Disorders (DSM-5) scale. This scale consists of 20 items on the symptoms of PTSD according to the DSM-5 criteria. Each item is rated from 0 ("not at all") to 4 ("extremely"). The maximum score is 80.
To define a predictive model of PTSD in this population | at 3 months after the patient's discharge from the ICU
  The primary endpoint is the proportion of family members who developed PTSD 3 months after the patient's discharge from the ICU assessed by the Post-traumatic stress disorder CheckList (PCL-5) version Diagnostic and Statistical Manual of Mental Disorders (DSM-5) scale. This scale consists of 20 items on the symptoms of PTSD according to the DSM-5 criteria. Each item is rated from 0 ("not at all") to 4 ("extremely"). The maximum score is 80.

SECONDARY OUTCOMES:
Assessing the psychological impact of a family member stay in intensive care | at inclusion, at the patient's discharge from the ICU, 3 and 6 months after the patient's discharge from the ICU
  Proportion of family members who developed symptoms of anxiety and depression assessed by the Hospital Anxiety and Depression Scale (HADS),
Assessing the psychological impact of a family member stay in intensive care | 6 months after the patient's discharge from the ICU
  Proportion of family members who developed PTSD 6 months after discharge from the assessed by the PCL-5 scale
Assessing the psychological impact of a family member stay in intensive care | at inclusion, at the patient's discharge from the ICU, 3 and 6 months after the patient's discharge from the ICU
  Proportion of relatives who developed severe insomnia assessed by the Insomnia Severity Index (ISI)
Assessing the psychological impact of a family member stay in intensive care | at inclusion, at the patient's discharge from the ICU, 3 and 6 months after the patient's discharge from the ICU
  Proportion of resilient relatives assessed by Resilience Scale (CD RISC 10)
Assessing the psychological impact of a family member stay in intensive care | at inclusion, at the patient's discharge from the ICU, 3 and 6 months after the patient's discharge from the ICU
  Proportion of relatives who developed peri-traumatic dissociation experiences (PDEQ)
Assessing the psychological impact of a family member stay in intensive care | at 6 months after the patient's death in intensive care
  Proportion of relatives who developed prolonged grief assessed by the Prolonged Grief disorder (PG-13) questionnaire
To identify the impact on the consumption of care and medical procedures of PTSD in family members of patients admitted to the ICU | at 3 and 6 months after discharge of the patient from the intensive care unit
  Proportion of relatives who used psychoactive substances assessed by the Who-assist questionnaire (Question 2 of the questionnaire), Consumption of care and medical procedures by relatives (MEDEC questionnaire

OTHER OUTCOMES:
Qualitative study | 3 to 4 months after the patient's death or discharge of the patient from the intensive care unit
  To deepen the understanding of the mechanisms leading to post-traumatic stress disorder in relatives of patients admitted to the ICU
  * Semi-structured interviews conducted by a psychologist or a sociologist
  * Population concerned by the interviews:
    1. relatives of non deceased patients (n= 20)
    2. bereaved relatives (patient who died in intensive care) (n= 20)
    3. nurses (n= 20) and intensive care physicians (n= 20).
FAME ICU Team (FIT) study | at the beginning of the study in the department
  to determine the individual and organizational (unit-related) factors associated with the risk of burnout among service professionals, and to identify a possible association between the presence of burnout and the ethical climate in which the professional working in the unit operates burnout and the ethical climate in which the professional working in the resuscitation.
  Scales completed by caregivers :
  * Maslach Burnout Inventory (MBI) for the assessment of burnout
  * Job Content Questionnaire (JCQ) for the assessment of job stress months").
  * Ethical Decision-Making Climate Questionnaire (EDMCQ) for the evaluation of the ethical climate
  * Professional Quality Of Life scale (ProQOL) for the assessment of quality of life at work
  * Connor-Davidson Resilience scale (CD-RISC 10) to assess resilience
  * Cultural Awareness Scale (CAS)
FAME Bio-bank: Analysis of molecular signatures of PTSD | to the inclusion
  The main objective is to provide a prediction of the risk of PTSD that is as close as possible to to the individuals concerned.

CONTACTS AND LOCATIONS:
Overall Officials: Jean REIGNIER, PU-PH, Principal Investigator — Nantes University Hospital
Locations (56):
- France (55):
  - CH Angoulême, Angoulême, France
  - Hôpital Privé d'Antony, Antony, France
  - CH d'Argenteuil, Argenteuil, France
  - CH de Bastia, Bastia, France
  - CH Beauvais, Beauvais, France
  - Hôpital Nord Franche Comté, Belfort, France
  - CH de Béthune, Beuvry, France
  - APHP Hôpital Avicenne, Bobigny, France
  - CHU de Bordeaux - Hôpital Saint-André, Bordeaux, France
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux, France
  - AP-HP Hôpital Ambroise Paré, Boulogne, France
  - CH de Boulogne-sur-Mer, Boulogne-sur-Mer, France
  - CHU de Brest, Brest, France
  - CH de Chartres, Chartres, France
  - CH de Cholet, Cholet, France
  - CHU Clermont-Ferrand - Centre Jean Perrin, Clermont-Ferrand, France
  - CHU Clermont-Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand, France
  - CH de Dieppe, Dieppe, France
  - CHU de Dijon, Dijon, France
  - CH de Fréjus - Saint Raphaël, Fréjus, France
  - APHP Hôpital Raymond Poincaré, Garches, France
  - CHU de Grenoble Alpes, Grenoble, France
  - GHEF- Site de Marne de la Vallée, Jossigny, France
  - CHD Vendée, La Roche-sur-Yon, France
  - CH de la Rochelle, La Rochelle, France
  - CH Versailles - Hôpital André Mignot, Le Chesnay, France
  - CH du Mans, Le Mans, France
  - CHU de Lille - Hôpital Roger Salengro, Lille, France
  - GHB Sud - Hôpital de Lorient, Lorient, France
  - CHU De Lyon - Hôpital Edouard Herriot, Lyon, France
  - AP-HM - Hôpital Nord, Marseille, France
  - Hôpital Privé Jacques Cartier, Massy, France
  - GHI le Raincy Montfermeil, Montfermeil, France
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier, France
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier, France
  - CHU de Nantes, Nantes, France
  - Clinique Ambroise Paré, Neuilly-sur-Seine, France
  - CHR d'Orléans, Orléans, France
  - APHP Hôpital Saint-Louis, Paris, France
  - APHP Hôpital Cochin, Paris, France
  - APHP Hôpital La Pitié Salpêtrière, Paris, France
  - APHP Hôpital Tenon, Paris, France
  - APHP Hôpital Saint-Antoine, Paris, France
  - CHI Poissy, Poissy, France
  - CH René Dubos, Pontoise, France
  - CH de Saint-Lô, Saint-Lô, France
  - CH de Saint-Nazaire, Saint-Nazaire, France
  - Hôpital du Pays Salonais, Salon-de-Provence, France
  - CH de Bassin de Thau, Sète, France
  - CH de Saint-Malo, St-Malo, France
  - Hôpital Foch, Suresnes, France
  - CH de Tourcoing - Hôpital Guy Chatiliez, Tourcoing, France
  - Ch Bretagne Atlantique - site de Vannes, Vannes, France
  - CH de Vichy, Vichy, France
  - Institut Gustave Roussy, Villejuif, France
- CHU La Guadeloupe, Pointe-à-Pitre, France, Guadeloupe